CLINICAL TRIAL: NCT03842735
Title: Promotion of Physical Activity for Children and Adolescents Undergoing Hematopoietic Stem Cells Transplantation (HSCT) During the In-patient Phase
Brief Title: Physical Activity in Children During Hematopoietic Stem Cells Transplantation (HSCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Francesca Rossi, Development Neuro and Psychomotor Therapist, A.O.U. Città della Salute e della Scienza
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PHYSICALACTIVITYHSCT0-18YSIPP
Record Dates: First submitted 2019-01-29; First posted 2019-02-15 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Hematopoietic Stem Cell Transplantation; Child; Adolescent
Keywords: Physiotherapy; Rehabilitation; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Eligible patients who provided consent were assigned to one of the two groups according to a "cluster time" selection model. The methodology was discussed and agreed with expert methodologists of the A.O.U. Città della Salute e della Scienza research group and based assignation to the two groups according to the time of hospitalization: EG enrollment May 2016-December 2016, March 2017-May 2017, November 2017-June 2018 and CG enrollment January 2017-February 2017, June 2017-October 2017, July 2018-August 2018.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise and rehabilitation counselling (Experimental): Subjects enrolled in exercise group make physical exercises and receive rehabilitative counselling indications
  Interventions: Other: exercise and rehabilitation counselling; Behavioral: rehabilitation counselling
- rehabilitation counselling (Other): Subjects enrolled in exercise group only receive rehabilitative counseling indications.
  Interventions: Behavioral: rehabilitation counselling

INTERVENTIONS:
Other: exercise and rehabilitation counselling — The intervention consists in a standardized physical exercise (PE) and rehabilitation counselling indications (RCI). PE is done 5 days/week (2 days in autonomy by the patient with parents support and 3 days supervised). Each session lasts 30 minutes and this is supervised by one therapist for all patients. Patients are enrolled in an EP composed by three different types of exercises, each carried out for 10 minutes per session: muscle strength exercises for upper and lower extremities preceded by warming up, aerobic exercises and stretching. The kind of exercise is differentiated by age range (children, 5-12 years and adolescents, 13-18 years).
  Other Names: rehabilitation
  Arms: exercise and rehabilitation counselling
Behavioral: rehabilitation counselling — RCI, which have to be followed daily, consist in some practical advice was given on how to adopt an active lifestyle during the recovery (e.g., getting up to go to the bathroom, getting up to move to the window to talk with visitors, sit on chair to have school lessons).

SUMMARY:
This interventional study was designed to assess the validity and the impact of a rehabilitation program on pediatric cancer patients undergoing hematopoietic stem cells transplantation (HSCT). Each participant will be randomly assigned to either an experimental or control (counseling rehabilitation care) group. The experimental group participate in an inpatient rehabilitation program for the duration of HSCT pathway. The program include standardized activities for 5 days a week in the child's room or in a pediatric gym at the hospital.

DETAILED DESCRIPTION:
BACKGROUND Hematopoietic stem cell transplantation (HSCT) is a potentially curative option for many diseases, such as hematologic malignancies and refractory solid tumors among children and adolescents. This procedure led to considerable improvement in survival rates, but also contributed to the development of late effects. Due to the severity of conditioning regimen, length of isolation and hospitalization period, weakness related to immunosuppression and drug toxicities, physical, cognitive and psychosocial functions are severely impaired. HSCT recipients may report impairments in cardiorespiratory fitness (fatigue), muscle bulk and strength, immunologic recovery, neuropsychological functions, functional abilities and autonomy with an undeniable decline of quality of life (QoL). Recently pediatric oncological research attentions have been directed to reduction of the impact of these side effects and to improvement of QoL, both during and after cancer treatment. The published studies about the effects of rehabilitation care, in pediatric population undergoing HSCT show how rehabilitation, which consists in structured and adapted different therapeutic activities, is safe and feasible. In particular studies conducted on the inpatient phase for HSCT report how the execution of a low intensity level of activity doesn't have any bad effect on immunological recovery, positively affects BMI, gives benefits on general health status, improves QoL, protects from depressive symptoms by promoting a healthy lifestyle during survivorship. Moderate exercise in a chronic graft-versus-host disease (cGVHD) murine model receiving total body irradiation (TBI) and immunosuppression can reduce clinical severity scores, blood interleukine-4 (IL-4) and tumor necrosis factor α levels while increasing survival, physical fitness, circulating B220 and cluster of differentiation 4 (CD4) lymphocytes. Finally, rehabilitation can improve immune function which has an impact on cancer control. Pediatric Oncohaematology Department of "Regina Margherita" Children's Hospital in Turin ["A.O.U. Città della Salute e della Scienza"] is one of the most important structure in Italy for pediatric HSCT. In the year 2016, 47 patients underwent HSCT: 25 of them were less than 11 years old and 22 were older than 11 years. In 2017, until the month of August, 25 patients were transplanted: 12 of them were less than 11 years old and 13 were older than 11 years. The in-patient phase lasted for a medium time of 40 days. From a recent review of the Department, in the period between March 2010 and November 2015, 207 children and adolescent patients benefited of a rehabilitation treatment, 42 of these during and after hospitalization for HSCT. However, to date rehabilitation programs have been implemented in a purely personalized perspective thus ignoring primary methodological issues (e.g., absence of a control group) which would allow an appropriate evaluation of outcomes generalizable to the target population. Therefore, rigorous interventions are mandatory in order to prevent future long-term treatment effects, to improve general health state of these patients and to share evidence-based guidelines for the optimal design for rehabilitation care in pediatric oncology.

EXPERIMENTAL PROJECT Starting from literature data on benefits of participation to a rehabilitation program for subjects undergoing HSCT, the current research intends to propose a project in a prevention perspective aim at the promotion of healthy life style for children and adolescents.

Procedures According to the difficulties reported in other studies that had both exercise group (EG) and control group (CG) patients recovery at the same time, and since this led to inevitable contamination between these two groups, investigators established that eligible patients who provided consent will be assigned to one of the two groups according to a "cluster time" selection model. The study it has been approved by the hospital's Ethical Committee. Written informed consent will be obtain from the participants or from their parents/guardians for patients under eighteen.

Exercise Intervention The study is presented to eligible patients and to their caregivers by a Development Neuro and Psychomotor Therapist in an interview. The interview regards: 1) problems that may occur during the HSCT procedure; 2) the importance of rehabilitation during the recovery to limit side effects; 3) presentation of the study design and procedures; 4) submission of the informed consensus. After having obtained the consensus, patients are assigned to the EG or the CG, according to the methodology previously explained. Subjects receive information booklets containing practical rehabilitation instructions, expressed in both text and illustrations, differentiated by the three identified age ranges (0-4, 5-12, 13-18). The content of booklets varies between EG and CG, since in the first case it contains both exercise and RCI, while for CG it regards only on RCI.

EXPERIMENTAL GROUP: The intervention consists in a standardized PE and RCI. PE is done 5 days/week (2 days in autonomy by the patient with parents support and 3 days supervised). Each session lasts 30 minutes and this is supervised by one therapist for all patients. Children aged less than 5 years make activities directed to sustain and promote their neuro-psychomotor development and muscle strength (e.g. to sit in the infant seat, playing in sitting position without support, playing on the floor and to crawl). Patients belonging to the other two age ranges are enrolled in an exercise programme (EP) composed by three different types of exercises, each carried out for 10 minutes per session: muscle strength exercises for upper and lower extremities preceded by warming up, aerobic exercises and stretching. For children aged 5-12 years activities are based principally on games (e.g. games with the ball, with circles and bricks, etc.), while structured exercises are proposed to adolescents (e.g. using weights, treadmills or exercise bikes); in both groups, the active videogames of Nintendo Wii(™) Fit is used to promote aerobic training. The EP is done only if the patient had platelets > 20000 and Hb > 8.0. Patients belonging to the upper age ranges also benefit from RCI, which has to be followed daily, and where some practical advice are given on how to adopt an active lifestyle during the recovery (e.g., getting up to go to the bathroom, getting up to move to the window to talk with visitors, sit on chair to have school lessons).

Parents record daily their child's EP and RCI activities in appropriate grids, and adolescents filled them in themselves.

CONTROL GROUP: Parents of children who belonged to the 0-4 years old age range CG receive a booklet with some RCI on how to reduce the time spent in bed and to propose different kinds of activities useful to sustain their development, according to the functional level of their child. Children who aged more than 5 years and adolescents of the CG receive the same part of the pamphlets given to the EG, containing written and illustrated indications of the RCI. The RCI has to be followed daily. Parents are required to record in appropriate grids their child's daily activities and adolescents filled them in themselves. The therapist goes 3 times/week to check that the diary has been filled in correctly.

EXPECTED RESULTS (experimental group vs control group): - Stable level of gross motor skills, functional motility, resistance to the walking and muscular strength from T0 and T1; - Stable level in passive articular movement in tibial artery dorsiflexion from T0 and T1; - Stable level of muscular elasticity from T0 and T1; - High perception of QoL and less fatigue from T0 and T1; - Improvement in immune functions; - Positive association between food intake and program participation.

FUTURE APPLICATIONS TO HEALTH The current project seeks to obtain not only important health and clinical benefits for patients undergoing HSCT in terms of late diseases reducing (e.g., obesity), but it will also underline new important association between exercise and biological system useful to find new insight for antitumor mechanisms. Also the need to improve several rehabilitation issues will be showed. For instance, the project will allow to focus on the importance that all patients have access to rehabilitation options. Actually, there is currently a gap between what investigators know from research, and what health care professionals, are implementing in pediatric cancer care. In Italy, for instance, the possibility to benefit of rehabilitation care is still poor because of the absence of services and facilities in several centres of pediatric oncology. So, to pay attention to these unmet needs will be the first step towards the reduction of the financial burden of hospitalization because of late effects problems and secondary disease some of which can be prevented with an appropriate rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* i) being children or adolescents (6 months -18 years old);
* ii) to have a diagnosis of oncological or hematological disease;
* iii) receiving an autologous or allogeneic HSCT;
* iv) to have spoken and written Italian language comprehension, both by children/adolescents and by parents.

Exclusion Criteria:

* i) to be affected by cognitive difficulties that preclude to the program's participation;
* ii) to be already undergoing rehabilitation before the entrance in the Transplantation Stem Cell Unit (TSCU).

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
change in global motor skills level | this outcome it is measured in the week before HSCT [Time 0] and post hematopoietic stem cells transplantation (HSCT), after the discharge from stem cells unit (SCU), at an average of 40 days after Time 0 [Time 1]
  The Gross Motor Function Measure (GMFM), version -88 for children who aged between 0-4 years, and version-Acute Lymphoblastic Leukemia (ALL) for older subjects. The GMFM-88 is composed by 88 items, while the GMFM-ALL is composed by 21 items. Each item can be scored as 0, 1, 2, 3, or "not tested". Scoring key: 0 - does not initiate, 1 - initiates, 2 - partially completes, and 3 - completed. The total score for GMFM-88 can be between 0 and 264, while for the GMFM-ALL can vary from 0 to 63.
change in range of passive ankle dorsiflexion | this outcome it is measured in the week before HSCT [Time 0] and post HSCT, after the discharge from SCU, at an average of 40 days after Time 0 [Time 1]
  Goniometer
rate of immune cells recovery | this outcome it is measured 35 days after the first day of infusion ("day zero")
  blood counts of leukocytes, monocytes, and lymphocytes and main lymphocyte subpopulations and dendritic cells
participation rate at the exercise program | 24 hours
  Parents are required to record in appropriate grids their child's daily activities and adolescents fill them in themselves. The therapist goes 3 times/week to check that the diary is filled in correctly. This outcome it is measured daily during the stay in the SCU.
adhesion rate to rehabilitative counselling indications | 24 hours
  Parents are required to record in appropriate grids their child's daily activities and adolescents fill them in themselves. The therapist goes 3 times/week to check that the diary is filled in correctly. This outcome it is measured daily during the stay in the SCU.

SECONDARY OUTCOMES:
change in functional motility level | this outcome it is measured in the week before HSCT [Time 0] and post HSCT, after the discharge from SCU, at an average of 40 days after Time 0 [Time 1]
  Time Up and Go Test (TUG); it is measured only in children who aged more than 5 years.
change in tibialis anterior and quadriceps muscles strength level | this outcome it is measured in the week before HSCT [Time 0] and post HSCT, after the discharge from SCU, at an average of 40 days after Time 0 [Time 1]
  Medical Research Council Scale (MRC). This method involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly:
  0 No muscle activation
  1. Trace muscle activation, such as a twitch, without achieving full range of motion
  2. Muscle activation with gravity eliminated, achieving full range of motion
  3. Muscle activation against gravity, full range of motion
  4. Muscle activation against some resistance, full range of motion
  5. Muscle activation against examiner's full resistance, full range of motion It is measured only in children who aged more than 5 years.
change in flexibility level of the lower back and hamstring muscles | this outcome it is measured in the week before HSCT [Time 0] and post HSCT, after the discharge from SCU, at an average of 40 days after Time 0 [Time 1]
  Seat and Reach Test; it is measured only in children who aged more than 5 years.
change in functional exercise capacity level | this outcome it is measured in the week before HSCT [Time 0] and post HSCT, after the discharge from SCU, at an average of 40 days after Time 0 [Time 1]
  Two Minute Walk Test; it is measured only in children who aged more than 5 years.
change in fatigue level | this outcome it is measured in the week before HSCT [Time 0] and post HSCT, after the discharge from SCU, at an average of 40 days after Time 0 [Time 1]
  PedsQL Multidimensional Fatigue Scale. The PedsQL is an interview where item Scaling is based on 5-point Likert scale from 0 (Never) to 4 (Almost always).Items are reversed scored and linearly transformed to a 0-100 scale as follows:
  0=100, 1=75, 2=50, 3=25, 4=0. Total Score: Sum of all the items over the number of items answered.
change of quality of life level: PedsQL Cancer Module | this outcome it is measured in the week before HSCT [Time 0] and post HSCT, after the discharge from SCU, at an average of 40 days after Time 0 [Time 1]
  PedsQL Cancer Module

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Rossi, Dr, Principal Investigator — A.O.U. Città della Salute e della Scienza - OIRM, Turin, Italy
Locations (1):
- A.O.U. Città della Salute e della Scienza - Regina Margherita children hospital, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossi F, Coppo M, Zucchetti G, Bazzano D, Ricci F, Vassallo E, Nesi F, Fagioli F. Rehabilitative intervention during and after pediatric hematopoietic stem cell transplantation: An analysis of the existing literature. Pediatr Blood Cancer. 2016 Nov;63(11):1895-904. doi: 10.1002/pbc.26114. Epub 2016 Jul 13. PMID 27409063
- [Background] Fiuza-Luces C, Soares-Miranda L, Gonzalez-Murillo A, Palacio JM, Colmenero I, Casco F, Melen GJ, Delmiro A, Moran M, Ramirez M, Lucia A. Exercise benefits in chronic graft versus host disease: a murine model study. Med Sci Sports Exerc. 2013 Sep;45(9):1703-11. doi: 10.1249/MSS.0b013e31828fa004. PMID 23954992
- [Background] Fiuza-Luces C, Gonzalez-Murillo A, Soares-Miranda L, Martinez Palacio J, Colmenero I, Casco F, Melen G, Moran M, Lucia A, Ramirez M. Effects of exercise interventions in graft-versus-host disease models. Cell Transplant. 2013;22(12):2409-20. doi: 10.3727/096368912X658746. Epub 2012 Oct 31. PMID 23127525
- [Background] Timmons BW, Cieslak T. Human natural killer cell subsets and acute exercise: a brief review. Exerc Immunol Rev. 2008;14:8-23. PMID 19203081
- [Background] Chamorro-Vina C, Ruiz JR, Santana-Sosa E, Gonzalez Vicent M, Madero L, Perez M, Fleck SJ, Perez A, Ramirez M, Lucia A. Exercise during hematopoietic stem cell transplant hospitalization in children. Med Sci Sports Exerc. 2010 Jun;42(6):1045-53. doi: 10.1249/MSS.0b013e3181c4dac1. PMID 19997035
- [Background] Rosenhagen A, Bernhorster M, Vogt L, Weiss B, Senn A, Arndt S, Siegler K, Jung M, Bader P, Banzer W. Implementation of structured physical activity in the pediatric stem cell transplantation. Klin Padiatr. 2011 May;223(3):147-51. doi: 10.1055/s-0031-1271782. Epub 2011 Apr 1. PMID 21462101
- [Background] Hayes S, Davies PS, Parker T, Bashford J, Newman B. Quality of life changes following peripheral blood stem cell transplantation and participation in a mixed-type, moderate-intensity, exercise program. Bone Marrow Transplant. 2004 Mar;33(5):553-8. doi: 10.1038/sj.bmt.1704378. PMID 14716346
- [Background] Chamorro-Vina C, Guilcher GM, Khan FM, Mazil K, Schulte F, Wurz A, Williamson T, Reimer RA, Culos-Reed SN. EXERCISE in pediatric autologous stem cell transplant patients: a randomized controlled trial protocol. BMC Cancer. 2012 Sep 10;12:401. doi: 10.1186/1471-2407-12-401. PMID 22963378
- [Background] Tanir MK, Kuguoglu S. Impact of exercise on lower activity levels in children with acute lymphoblastic leukemia: a randomized controlled trial from Turkey. Rehabil Nurs. 2013 Jan-Feb;38(1):48-59. doi: 10.1002/rnj.58. Epub 2012 Oct 18. PMID 23365005
- [Background] Hartman A, Hop W, Takken T, Pieters R, van den Heuvel-Eibrink M. Motor performance and functional exercise capacity in survivors of pediatric acute lymphoblastic leukemia. Pediatr Blood Cancer. 2013 Mar;60(3):494-9. doi: 10.1002/pbc.24243. Epub 2012 Jun 28. PMID 22745035
- [Background] Moyer-Mileur LJ, Ransdell L, Bruggers CS. Fitness of children with standard-risk acute lymphoblastic leukemia during maintenance therapy: response to a home-based exercise and nutrition program. J Pediatr Hematol Oncol. 2009 Apr;31(4):259-66. doi: 10.1097/MPH.0b013e3181978fd4. PMID 19346877
- [Background] Braam KI, van der Torre P, Takken T, Veening MA, van Dulmen-den Broeder E, Kaspers GJ. Physical exercise training interventions for children and young adults during and after treatment for childhood cancer. Cochrane Database Syst Rev. 2016 Mar 31;3(3):CD008796. doi: 10.1002/14651858.CD008796.pub3. PMID 27030386
- [Derived] Rossi F, Zucchetti G, Esposito M, Berchialla P, Sciannameo V, Vassallo E, Saglio F, Chamorro Vina C, Scarrone S, Vittorini R, Fagioli F. Rehabilitation in children and adolescents undergoing stem cell transplantation: A pilot study focused on motor performance. Eur J Cancer Care (Engl). 2022 Nov;31(6):e13711. doi: 10.1111/ecc.13711. Epub 2022 Sep 28. PMID 36168857